CLINICAL TRIAL: NCT02907320
Title: EXPLORATORY ASSESSMENT OF THE EFFECTS OF CYCLO 3 ® FORT (Ruscus Extract, Hesperidin Methyl Chalcone, Ascorbic Acid) OR MICRONISED PURIFIED FLAVONOID FRACTION ON VASCULAR PARAMETERS AND BIOMARKERS IN WOMEN SUFFERING FROM CHRONIC VENOUS DISEASE (CEAP C2 OR C3), OVER 8 WEEKS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Eurotrials Brasil Consultores Cientificos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DC0982 GE 2 04
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Venous Disease Classification (CEAP): C2 or C3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CYCLO 3 ® FORT and placebo MPFF (Experimental): MPFF = Micronized Purified Flavonoid Fraction
  Interventions: Drug: CYCLO 3 ® FORT; Drug: placebo MPFF
- MPFF and placebo CYCLO 3 ® FORT (Active Comparator): MPFF = Micronized Purified Flavonoid Fraction
  Interventions: Drug: MPFF; Drug: placebo CYCLO 3 ® FORT
- placebo (Placebo Comparator): MPFF = Micronized Purified Flavonoid Fraction
  Interventions: Drug: placebo CYCLO 3 ® FORT; Drug: placebo MPFF

INTERVENTIONS:
Drug: CYCLO 3 ® FORT
  Arms: CYCLO 3 ® FORT and placebo MPFF
Drug: MPFF
  Arms: MPFF and placebo CYCLO 3 ® FORT
Drug: placebo CYCLO 3 ® FORT
  Arms: MPFF and placebo CYCLO 3 ® FORT; placebo
Drug: placebo MPFF
  Arms: CYCLO 3 ® FORT and placebo MPFF; placebo

SUMMARY:
Chronic Venous Disorder is the most prevalent vascular disease. It is multifactorial pathology that has an important impact on quality of life and represents a significant public health concern, due to its very high frequency in all European and American (north and south) countries.

Venous pathology develops when venous pressure is increased and return of blood is impaired through several mechanisms. Wish induce leg symptoms (tingling, aching, burning, pain, muscle cramps, sensation of swelling, sensations of throbbing or heaviness, itching skin, restless legs, leg tiredness and/or fatigue.

The aims of this research is to study the effects on microcirculatory activity (activity on very small vessels) of CYCLO 3 ® FORT, MPFF (Micronised Purified Flavonoid Fraction) and Placebo after 8 week of treatment by Microscan, and Duplex, two imaging non-invasive technologies will be performed to obtain measurements of microcirculatory parameters in standardized and reproducible conditions for all the participants. In addition, will assess, in blood samples, the inflammatory biomarkers .

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria

   * Non-menopausal women aged from 18 to 50 years
   * Symptomatic Primary chronic disorder C2 or C3 of advanced CEAP
   * Regular menstrual cycle
   * Use an efficient method of contraception
   * Having signed her written informed
2. Non-inclusion criteria 2.1 Related to pathology:

   * Superficial and or deep venous thrombosis
   * Venous insufficiency including history of deep venous thrombosis, post thrombotic syndrome, venous dysplasia, compressive syndrome
   * History of venous strapping or phlebotomy/ surgery of the evaluated leg
   * Sclerosing injection within 6 month before inclusion
   * Oedema from other etiology
   * Paresthesia, cramps of the lower limbs from other origin 2.2 Related to treatment:
   * Hypersensitivity, allergy or intolerance to study drugs
   * Iron storage disorder
   * Intake of venotonic treatment (oral or topic) ,triptan ,diuretics ,calcium blockers, beta blockers, ACE inhibitors, angiotensine II inhibitors, vasodilatators and/or vasoconstrictors within 1 month before inclusion
   * Intake of NSAID,corticosteroids,ergotamine, dihydroergotamine or any ergot alkaloids,vitamin C nutraceutical or phytotherapy products with potential venotonic effect within 2 weeks before inclusion 2.3 Related to the population:
   * History of diabetes
   * BMI≥ 30
   * Grade V and VI on Fitzpatrick classification

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change of Capillary diameter | From baseline (Day 0) to Day 56
  Measure by microscan of capillary diameter, in micrometer on the worst leg (CEAP classification C2 or C3) at Baseline.

SECONDARY OUTCOMES:
Change of venoconstriction activity | From baseline (Day 0) to Day 56
  Measure by Duplex-scan of vein diameter in millimeter on the worst leg (CEAP classification C2 or C3) at Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zahida Issiakhem Belkaid, MD, Study Director — Pierre Fabre Medicament

IPD SHARING:
Plan to Share IPD: No